CLINICAL TRIAL: NCT07211685
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Phase 2a Study With an Extension Phase to Evaluate the Efficacy and Safety of BAY 3401016 in Participants Aged 18 to 45 With Alport Syndrome
Brief Title: BAY3401016; Biomarker Study Alport
Acronym: ASSESS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22419
Record Dates: First submitted 2025-09-19; First posted 2025-10-08 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary

STUDY DESIGN:
Intervention Model Description: Two parallel groups (BAY 3401016 and placebo)
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAY 3401016 (Experimental): BAY 3401016 weekly for 24 weeks in addition to background therapy if eligible
  Interventions: Biological: BAY 3401016
- Placebo (Placebo Comparator): Placebo weekly for 24 weeks in addition to background therapy if eligible
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BAY 3401016 — BAY 3401016
  Arms: BAY 3401016
Other: Placebo — Placebo to BAY 3401016
  Arms: Placebo

SUMMARY:
Alport syndrome (AS) is a rare genetic condition that causes kidney disease, hearing loss, and eye abnormalities that occur due to changes in specific genes (COL4A3, COL4A4, and COL4A5). These genes help in producing an important protein called collagen. People with AS have a high risk of developing chronic kidney disease (CKD), a condition in which there is progressive loss in kidney function over time. The kidneys soon lose their ability to remove waste products from the body properly, resulting in end-stage kidney disease. A common sign of decreasing kidney function is the presence of excess protein in the urine that is not usually found with healthy kidneys. This condition is known as proteinuria. The study drug, BAY 3401016 (a monoclonal antibody), is a type of medicine that blocks a protein called Semaphorin 3A (Sema3A), which is thought to be involved in causing kidney damage in AS. By blocking the action of the Sema3A protein, BAY 3401016 may prevent proteinuria and slow down the loss in kidney function due to AS.

The main purpose of this study is to learn more about how well BAY 3401016 works in slowing down the loss in kidney function in adults with a rapidly progressing AS.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 45 years of age inclusive
* Participants with AS, either XLAS (male) or ARAS (male or female)
* eGFR ≥ 45 mL/min/1.73m2
* UACR ≥ 500mg/g

Exclusion Criteria:

* Chronic kidney disease is different from AS
* Clinically significant illness that could have influence on the safety of the participant and/or interfere with the study objectives
* History or current existence of malignancy
* Participants with history of severe allergies, multiple drug allergies or non-allergic drug reactions including allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids or urticaria
* Participants with active skin disorders (e.g. atopic dermatitis, severe acne)
* Systolic blood pressure above 140 mmHg
* Diastolic blood pressure above 90 mmHg

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2028-07-27 (Estimated); Study Completion 2028-07-27 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin creatinine ratio (UACR) ratio to baseline averaged over 16, 20 and 24 weeks of treatment | From the start of study intervention, over 16, 20 and 24 weeks of treatment, until the last follow-up visit, 90 days ± 3 days after EoT
  Progression of kidney disease, including Alport Syndrome (AS), to End-Stage Renal Disease (ESRD) takes years, making it challenging to establish drug efficacy in clinical trials without long follow-ups or large sample sizes. Using surrogate endpoints, such as early changes in albuminuria, can help address this issue. It is tested wether BAY 3401016 has an effect on albuminuria in AS patients. Research shows that albumin overload leads to renal function decline and podocyte injury.

SECONDARY OUTCOMES:
Investigate the safety and tolerability of BAY 3401016 in participants with AS | From the start of study intervention until the last follow-up visit, 90 days ± 3 days after EoT
  Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (6):
  - Nephrology Clinic at The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - The Peggy and Harold Katz Family Drug Discovery Center - Nephrology, Miami, Florida
  - Center for Advanced Pediatrics - Nephrology, Atlanta, Georgia
  - Cardio Renal Institute, Chubbuck, Idaho
  - Tufts Medical Center | Nephrology Department, Boston, Massachusetts
  - Renal Disease Research Institute | Landry, Dallas, Texas
- Argentina (4):
  - Hospital Británico, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro de Educacion Medica e Investigaciones Clinicas "Norberto Quirno" (CEMIC), Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro de Rehabilitacion Cardiovascular | San Luis, Argentina, San Luis, San Luis Province
  - Clinica de Nefrologia, Urologia y Enfermedades Cardiovasculares S.A., Santa Fe
- Canada (5):
  - St. Joseph's Healthcare - Hamilton, Hamilton, Ontario
  - London Health Sciences Centre (LHSC) - University Hospital, London, Ontario
  - Lakeridge Health-Oshawa, Oshawa, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
- China (5):
  - Peking University First Hospital - Department of Pediatrics, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University - Department of Nephrology, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University - Department of Pediatrics, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology - Pediatric Nephrology and Immunology, Wuhan, Hubei
  - Children's Hospital, Zhejiang University School of Medicine - Department of Nephrology, Hangzhou, Zhejiang
- Czechia (2):
  - Fakultní nemocnice Hradec Kralové - Nefrologická klinika, Hradec Králové
  - Všeobecná fakultní nemocnice v Praze - Klinika nefrologie, Prague
- France (4):
  - CHU bordeaux - Hopital Pellegrin - Service de Nephrologie-Transplantation-Dialyse-Aphereses, Bordeaux
  - CHU de Brest - Hopital La Cavale Blanche - Service de Nephorologie-Hémodialyse-Transplantation, Brest
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Necker-Enfants Malades - Service d'Hopital De Jour Néphrologie adulte, Paris
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital de Rangueil - Nephrologie et transplantation d'organes, Toulouse
- Germany (4):
  - Universitaetsmedizin Goettingen (UMG) - Klinik fuer Nephrologie und Rheumatologie, Göttingen, Lower Saxony
  - Universitaetsklinikum Koeln - Klinik II fuer Innere Medizin - Nephrologie, Rheumatologie, Diabetologie, Innere Medizin, Cologne, North Rhine-Westphalia
  - Charité Mitte - Nephrologie und Internistische Intensivmedizin, Berlin
  - Universitaetsklinikum Erlangen - Medizinische Klinik 4, Nephrologie, Hypertensiologie, Erlangen
- India (4):
  - Mavani Research Center, Ahmedabad, Gujarat
  - K.G. Hospital, Coimbatore
  - The Institute of Post Graduate Medical Education & Research (IPGMER) (SSKM Hospital), Kolkata
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi
- Italy (4):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Nefrologia, Dialisi e Trapianto, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia - Nefrologia, Brescia
  - IRCCS Istituto Giannina Gaslini - Nefrologia e Trapianto Rene, Genova
  - Ospedale Pediatrico Bambino Gesù - Nefrologia, Roma
- Japan (4):
  - Japanese RedCross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Saitama Prefectural Children's Medical Center, Chuo-Ku, Saitama
  - Kobe University Hospital, Kobe
  - Local Incorporated Administrative Agency Osaka City Hospital Organization Osaka City General Hospital, Osaka
- Poland (3):
  - CSK U.M. Lodz - Klin. Nefrologii, Hipertensjologii, Transplantologii i Chorób Wewnetrznych Samodz. Publiczny Zaklad OZ, Lodz
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Oddzial Kliniczny Nefrologii Transplantologii i Chorob Wewnetrznych, Poznan
  - Wojskowy Instytut Medyczny Panstwowy Instytut Badawczy - Centrum Wsparcia Badan Klinicznych, Warsaw
- Portugal (4):
  - Hospital de Curry Cabral - Nephrology Department, Lisbon
  - ULS São João - Nephrology Department, Porto
  - Hospital de Torres Novas - Nephrology Department, Torres Novas
  - Unidade Local de Saude de Gaia/Espinho E.P.E Nephrology Department, Vila Nova de Gaia
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (5):
  - Hospital La Mancha Centro_Nephrology, Alcázar de San Juan, Ciudad Real
  - Hospital Universitari Vall d´Hebron_ Nefrologia, Barcelona
  - Fundació Puigvert Enfermedades Renales Hereditarias. Servicio de Nefrología, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz | Nephrology and Hypertension Department, Madrid
  - Hospital Universitario Virgen del Rocio_Nephrology, Seville
- United Kingdom (4):
  - South Tyneside and Sunderland NHS Foundation Trust | Sunderland Royal Hospital - Renal Unit, Sunderland, Tyne and Wear
  - Royal Devon University Healthcare NHS Foundation Trust | Royal Devon and Exeter Hospital - Renal Unit, Exeter
  - Royal Free London NHS Foundation Trust | Royal Free Hospital - Centre for Nephrology, London
  - Sheffield Teaching Hospitals NHS Foundation Trust | Northern General Hospital - Sheffield Kidney Institute, Sheffield

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.